CLINICAL TRIAL: NCT03393429
Title: Training Therapy for the Secondary and Tertiary Prevention of Backache and Low Back Pain: A Randomized Controlled Pilot Study
Brief Title: Training Therapy for the Prevention of Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Gerold Ebenbichler, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1118/2012
Record Dates: First submitted 2018-01-03; First posted 2018-01-08 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Back Pain; Lower Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAVID assisted training (Active Comparator): Group I: Training assisted by DAVID devices
  Interventions: Other: DAVID assisted training
- training recommendation (Placebo Comparator): Group II: Training based on "stay active" recommendations
  Interventions: Other: training recommendation

INTERVENTIONS:
Other: DAVID assisted training — DAVID device assisted training under supervision
  Arms: DAVID assisted training
Other: training recommendation — training recommendation to "stay active"
  Arms: training recommendation

SUMMARY:
Work place related (lower) back pain in medical personnel is limiting to workability.

Even though occupational prevention programs are increasingly established, data on the effectiveness of training interventions offered at work-sites is largely missing.

In this randomized, investigator-blind, controlled feasibility study we aim to compare the effectiveness of device assisted training therapy in comparison to a general recommendation "to stay active" or group gymnastics in terms of pain frequency and intensity (main outcome). Additional outcome variables are: quality of life, psychological well-being, work efficiency, of sick-leave days.

Eligible employees (2 x 30) of the General Hospital of Vienna (AKH) over the age of 45 years suffering from (lower) back pain (>30 days/last year) of intensity ≥ 3 (numeric scale 0-10) will be included in two parallel groups. Group I starts with a device (DAVID) assisted training (40 training sessions; 2x / week) of the core trunk musculature. Group II gets instructions and an advice on how to "stay active" during the first 6 months. Assessment will be conducted before and after these 6 months; then groups are switched, thus, study subjects act as their own controls.

DETAILED DESCRIPTION:
Work place related pain syndromes of the (lower) back pose a major health problem for medical personnel. Beside the discomfort and limitations of the affected patients, a severe restriction of their ability to work must be considered.

For secondary prevention of back pain, health promotion programs are recommended. These consist of psychosocial and ergonomic interventions and, above all, a regular strengthening of the stabilizing muscle groups. Specific strength and endurance training for the trunk musculature with appropriate equipment is considered as a useful preventive measure and thus commonly offered at large corporations, even during working hours of the staff. However, data clearly demonstrating the effectivity and cost-effectiveness of these interventions is largely missing.

This pilot study serves several purposes:

On one hand, the feasibility of a randomized, controlled study is to be examined, which is to prove the effectiveness of the medical training therapy in comparison to a general recommendation "to stay active" or in comparison to group gymnastics. In particular, logistical problems in the organization of training therapy and training compliance must be clarified.

On the other hand, this pilot study serves to generate hypotheses. Several variables in regard to possible changes due to the training intervention will be investigated. Collected pilot data will be used for corresponding case number estimates of a subsequent confirmatory study. The outcome variables are: number of back pain days and intensity, quality of life, psychological well-being, work efficiency, days of sick-leave.

Study Design Randomized, investigator-blind, controlled pilot study with parallel group comparison of outcomes in employees of the General Hospital of Vienna (AKH) over the age of 45 years

Study Subjects 2 x 30 employees over the age of 45, who suffered more than 30 days of back and / or lower back pain of moderate to high intensity ≥ 3 (numeric scale 0-10) in the last year and suffer from pain in up to 3 body parts (in total) or less. Group I starts with a machine assisted training, group II starts after a period of observation half a year later.

Study Interventions 40 training sessions (2x / week) with DAVID training machines, which aim to improve the strength, endurance and performance of the core trunk musculature. The training will be initiated after a sufficiently long period of adjustment to the guidelines of the American College of Sports Medicine. The training plan is created individually for each subject. 4 to 6 people per hour can work out simultaneously. The training should be completed in max 6 months or less.

Group II gets instructions and an advice on how to "stay active" during the first 6 months. Assessment will be conducted before and after these 6 months.

After 6 months the groups are switched (group I with the initial DAVID machine assisted training is left with recommendations to "stay active"; subjects from group II are now trained for 6 months by means of 40 training sessions (2x / week) with DAVID assistance), thus, study subjects act as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* subjects must have suffered from (low) back pain for at least 6 days in the last month, without treatment by a doctor or feeling in need of treatment.
* subject reported pain should reach the level of 3 or more on the numeric rating scale of 0-10 (0 equals no pain and 10 represents the strongest imaginable pain) [Larsen et al, 2008; Blagsted et al., 2008].
* protocol documenting pain and work disability/limitations daily for a month must be completed
* written consent after completed patient education by a physician must be given

Exclusion Criteria: (one or more of the following)

* in order to rule out generalized musculoskeletal disorders, subjects should report discomfort or pain in no more than 3 different body parts
* arterial hypertension and cardiovascular events such as myocardial infarction within the last year and / or cardiomyopathy NYHA III and IV.
* symptomatic, lumbar disc herniation with associated neurological deficits
* specific spinal diseases as potential underlying reason for a back pain syndrome including rheumatoid arthritis, ankylosing spondylitis, manifested osteoporosis with St.p. vertebral fractures, tumors.
* St.p. traumatic damage of spine, pelvis or femur in the last 6 months
* insufficiently healed surgical wounds in any body area
* imminent musculoskeletal, spinal, hip or knee surgery
* chronic infectious diseases
* diagnosed mental illness
* previous severe trauma with permanent Musculoskeletal dysfunction
* pregnancy prior to study entrance examination
* no written consent to the study
* less than 1 year before retirement or planned job change within one year

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Frequency | 6 months
  Incidence of pain-days and pain-intensity

SECONDARY OUTCOMES:
Sick-Leave | 6 months
  Days of sick-leave in total

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Ebenbichler, Prof. Dr., Principal Investigator — University Department of Physical Medicine, Rehabilitation and Occupational Medicine
Locations (1):
- University Department of Physical Medicine, Rehabilitation and Occupational Medicine, Vienna, Austria